CLINICAL TRIAL: NCT01573416
Title: "Effectiveness of a Brief Intervention for Substances Consumption Linked to the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST): A Randomized Control Trial in Chilean Primary Care."
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Servicio Nacional para la Prevención y Rehabilitación del Consumo de Drogas y Alcohol (SENDA) (Unknown)
Responsible Party: Principal Investigator, Fernando Poblete Arrué, Profesor Asistente Adjunto, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEDAUC-11-205
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2012-04

CONDITIONS: Alcohol-Related Disorders; Substance-Related Disorders; Substance Abuse
Keywords: Alcohol; Abuse; Drugs; Brief intervention; ASSIST
MeSH Terms: conditions — Alcohol-Related Disorders; Substance-Related Disorders; Helping Behavior | interventions — Observation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Placebo Comparator)
  Interventions: Other: Observation
- Intervention group (Active Comparator)
  Interventions: Other: ASSIST-linked brief intervention for hazardous and harmful substance use.

INTERVENTIONS:
Other: ASSIST-linked brief intervention for hazardous and harmful substance use. — ASSIST-linked brief intervention will be applied to users achieving moderate risk scores in the ASSIST questionnaire. If after randomization are selected to enter the intervention group, they will receive a ten minute counseling carried immediately after the screening instrument. This intervention group will be re-evaluated after 3 months with the same ASSIST screening instrument.
  Arms: Intervention group
Other: Observation — Subjects who obtain a moderate risk score in the ASSIST screening questionnaire and after randomization are selected for the control group, will receive a brochure with substance-abuse information without any further conversation about the subject with the caregiver. This observation group will be re-evaluated after 3 months with the same ASSIST screening instrument.
  Arms: Control group

SUMMARY:
Alcohol and drugs consumption are among the highest risk factor for health in Chile and abroad. In Chile, harmful use of alcohol continues to be a major contributor to the burden of disease while lost years of healthy life are higher than many other risk factors such as hypertension, overweight and obesity, and hyperglycemia. It is important to say that the impact of alcohol consumption is greater in younger age groups where fatal injuries occur relatively early in life, as well.

In Chile, the consumption pattern in 2008 showed that 49.8 % consumed at least once in the last month for alcohol, 3.5 % for marihuana and 1.3 % for cocaine. This prevalence was even greater in young adults and adolescents and is associated with other mental health issues and poorer life quality. Those who have consumed marihuana during the last year, 25% report dependence symptoms. For cocaine derives, dependency rises up to 50% among the consumers. This data reinforce the need to design and implement strategies for reducing alcohol and drugs consumption in our population.

Also, it is well known that a high number of those who suffers from any addiction problem do not get attention in a specialized center. The are many barriers to do so, such as lack of motivation, lack of resources, social problems, access to care problems, and so on.

Chile has a shortage of preventive interventions for those at risk to develop an addiction at an early stage of substance use because front line health services (Primary health care and emergency care) and other social services (police stations, local justice courts) do not have a screening system and a model of brief intervention.

The Pontificia Universidad Catolica de Chile, through its Addiction Studies Center (CEDA UC) and its Department of Family Medicine, is working in conjunction with SENDA (Servicio Nacional para la Prevención y Rehabilitación del Consumo de Drogas y Alcohol ) to design, implement and evaluate a communal system for early detection, brief intervention and referral to treatment (SBIRT), in people older than 18 years, with substance consumption in five municipalities in the country.

The aid of this study is to demonstrate that a model of brief intervention is more effective than the approach currently used in patients with substance use at moderate risk (i.e.follow-up). It is a multicentric randomized controlled trial, single blind, with a group to receive brief intervention and a control group that is kept in control and waiting list being re-evaluated three months later.

The target population is composed by users whose ASSIST screening scores place them in the moderate risk group, for which there has not been defined a structured intervention yet by our health system. The information will be obtained from the scores obtained after the application of the ASSIST-WHO questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 18 years and 50 years
* Achieving a moderate risk score in the ASSIST screening questionnaire.
* Without any similar intervention in the last 3 months. (ie. AUDIT test).

Exclusion Criteria:

* Pregnant women.
* Users with cognitive disabilities.
* Users with language and communication disabilities.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Post-intervention ASSIST screening score. | 3 months
  3 months after being recruited, users with moderate risk in the ASSIST questionnaire who received either a brief intervention or observation will be re-evaluated with the same ASSIST instrument. In both the intervened and the control group, changes in the post-intervention ASSIST score will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Poblete, MD, MPH, Study Director — Pontificia Universidad Catolica de Chile
Locations (30):
- Chile (30):
  - CESFAM Dr. Sergio Aguilar, Coquimbo, IV
  - CESFAM San Juan, Coquimbo, IV
  - CESFAM Santa Cecilia, Coquimbo, IV
  - CESFAM Tierras Blancas, Coquimbo, IV
  - SAPU Dr. Sergio Aguilar, Coquimbo, IV
  - SAPU Tierras Blancas, Coquimbo, IV
  - 5ta. Comisaría Conchalí, Conchalí, RM
  - CS Alberto Bachelet, Conchalí, RM
  - CS José Symon Ojeda, Conchalí, RM
  - CS Juanita Aguirre, Conchalí, RM
  - CS Lucas Sierra, Conchalí, RM
  - SAPU Lucas Sierra, Conchalí, RM
  - 43va. Comisaría Peñalolén, Peñalolén, RM
  - CESFAM Lo Hermida, Peñalolén, RM
  - CESFAM Padre Gerardo Whelan, Peñalolén, RM
  - CS Carol Urzúa Ibañez, Peñalolén, RM
  - CS La Faena, Peñalolén, RM
  - SAPU Lo Hermida, Peñalolén, RM
  - 26va. Comisaría Pudahuel, Pudahuel, RM
  - CESFAM Gustavo Molina, Pudahuel, RM
  - CESFAM RAúl Silva Henríquez, Pudahuel, RM
  - CESFAM Violeta Parra, Pudahuel, RM
  - Consultorio Estrella, Pudahuel, RM
  - SAPU La Estrella, Pudahuel, RM
  - 14va. Comisaría San Bernardo, San Bernardo, RM
  - APS Carol Urzúa, San Bernardo, RM
  - APS Confraternidad, San Bernardo, RM
  - APS El Manzano, San Bernardo, RM
  - APS Raúl Cuevas, San Bernardo, RM
  - SAPU Raúl Brañes, San Bernardo, RM

REFERENCES:
- [Background] Humeniuk R, Ali R, Babor T, Souza-Formigoni ML, de Lacerda RB, Ling W, McRee B, Newcombe D, Pal H, Poznyak V, Simon S, Vendetti J. A randomized controlled trial of a brief intervention for illicit drugs linked to the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) in clients recruited from primary health-care settings in four countries. Addiction. 2012 May;107(5):957-66. doi: 10.1111/j.1360-0443.2011.03740.x. Epub 2012 Feb 28. PMID 22126102
- [Background] Beich A, Thorsen T, Rollnick S. Screening in brief intervention trials targeting excessive drinkers in general practice: systematic review and meta-analysis. BMJ. 2003 Sep 6;327(7414):536-42. doi: 10.1136/bmj.327.7414.536. PMID 12958114
- [Background] Ballesteros J, Duffy JC, Querejeta I, Arino J, Gonzalez-Pinto A. Efficacy of brief interventions for hazardous drinkers in primary care: systematic review and meta-analyses. Alcohol Clin Exp Res. 2004 Apr;28(4):608-18. doi: 10.1097/01.alc.0000122106.84718.67. PMID 15100612
- [Background] Hungerford DW, Pollock DA, Todd KH. Acceptability of emergency department-based screening and brief intervention for alcohol problems. Acad Emerg Med. 2000 Dec;7(12):1383-92. doi: 10.1111/j.1553-2712.2000.tb00496.x. PMID 11099429
- [Background] Anderson PA, Grey SF, Nichols C, Parran TV Jr, Graham AV. Is screening and brief advice for problem drinkers by clergy feasible? A survey of clergy. J Drug Educ. 2004;34(1):33-40. doi: 10.2190/3QH2-VLWN-ELWM-KC67. PMID 15468746
- [Background] Babor TF, McRee BG, Kassebaum PA, Grimaldi PL, Ahmed K, Bray J. Screening, Brief Intervention, and Referral to Treatment (SBIRT): toward a public health approach to the management of substance abuse. Subst Abus. 2007;28(3):7-30. doi: 10.1300/J465v28n03_03. PMID 18077300
- [Background] Gentilello LM, Rivara FP, Donovan DM, Jurkovich GJ, Daranciang E, Dunn CW, Villaveces A, Copass M, Ries RR. Alcohol interventions in a trauma center as a means of reducing the risk of injury recurrence. Ann Surg. 1999 Oct;230(4):473-80; discussion 480-3. doi: 10.1097/00000658-199910000-00003. PMID 10522717
- [Background] Babor TF, Kadden RM. Screening and interventions for alcohol and drug problems in medical settings: what works? J Trauma. 2005 Sep;59(3 Suppl):S80-7; discussion S94-100. doi: 10.1097/01.ta.0000174664.88603.21. PMID 16355071
- [Background] WHO ASSIST Working Group. The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST): development, reliability and feasibility. Addiction. 2002 Sep;97(9):1183-94. doi: 10.1046/j.1360-0443.2002.00185.x. PMID 12199834
- [Background] Whitlock EP, Polen MR, Green CA, Orleans T, Klein J; U.S. Preventive Services Task Force. Behavioral counseling interventions in primary care to reduce risky/harmful alcohol use by adults: a summary of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2004 Apr 6;140(7):557-68. doi: 10.7326/0003-4819-140-7-200404060-00017. PMID 15068985
- [Background] Hawks D. Broadening the base of treatment for alcohol problems: a report which deserves to be debated. The limits of treatment and importance of prevention. Br J Addict. 1991 Jul;86(7):848-9. doi: 10.1111/j.1360-0443.1991.tb01836.x. No abstract available. PMID 1912733
- [Derived] Greene MC, Kane J, Alto M, Giusto A, Lovero K, Stockton M, McClendon J, Nicholson T, Wainberg ML, Johnson RM, Tol WA. Psychosocial and pharmacologic interventions to reduce harmful alcohol use in low- and middle-income countries. Cochrane Database Syst Rev. 2023 May 9;5(5):CD013350. doi: 10.1002/14651858.CD013350.pub2. PMID 37158538
- See also: Pontificia Universidad Católica de Chile, School of Medicine — http://medicina.uc.cl
- See also: Servicio Nacional para la Prevención y Rehabilitación del Consumo de Drogas y Alcohol (SENDA) — http://www.senda.gob.cl
- See also: Family Medicine Dept., Pontificia Universidad Católica de Chile, School of Medicine. — http://medicinafamiliar.uc.cl